CLINICAL TRIAL: NCT06982677
Title: Improving Outcomes for Women Experiencing Premature or Early Menopause After Cancer: Development and Pilot Testing of a Novel Intervention
Brief Title: Improving Outcomes in Early Menopause After Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00117811
Record Dates: First submitted 2025-05-05; First posted 2025-05-21 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Early Menopause; Cancer
MeSH Terms: conditions — Primary Ovarian Insufficiency; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Behavioral Intervention (Experimental): Participants will engage in a 6-session program, to be delivered by a nurse navigator in an individual therapy setting, via telehealth. The program will integrate education, decision support, patient activation strategies, and cognitive-behavioral menopause symptom management skills.
  Interventions: Behavioral: Nurse Navigator Intervention
- Education Control (Other): Participants will receive the National Cancer Institute booklet, "Facing Forward: Life After Cancer Treatment," which provides basic strategies for navigating cancer survivorship.
  Interventions: Other: Education Control

INTERVENTIONS:
Behavioral: Nurse Navigator Intervention — The intervention will integrate education, decision support, patient activation strategies, and cognitive-behavioral menopause symptom management skills. Participants will receive video and audio-recorded materials and a written manual.
  Arms: Behavioral Intervention
Other: Education Control — The control arm will receive the National Cancer Institute booklet, "Facing Forward: Life After Cancer Treatment," which provides basic strategies for navigating cancer survivorship.
  Arms: Education Control

SUMMARY:
The goal of this study is to create and test a new program led by nurse navigators to help women who experience early menopause after cancer. The program includes personalized menopause education, decision support, and skills to manage menopause symptoms.

The main questions it aims to answer are:

1. Is the program easy to join, engaging, and well-received by participants?
2. Does the program group show greater improvements in knowledge, decision-making, confidence, and menopause symptom management compared to the control group?

Participants will complete sessions of either the program being tested or an educational control program with a nurse navigator via video. Participants will also complete questionnaires when they start the study and again about 10 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* female (biological sex);
* 18 to 44 years old;
* completed cancer treatment (other than endocrine therapy) >12 months prior to enrollment;
* have not had a period for more than 12 months (amenorrhea);
* able to speak and read English.

Exclusion Criteria:

* diagnosis of metastatic cancer;
* visual or hearing impairment that would interfere with participation in study;
* cognitive impairment or severe mental illness that would interfere with participation in study.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Enrollment | 10 months
  Feasibility will be assessed by examining trial enrollment over the course of 10 months. The trial will be considered feasible if the study enrolls N=60 participants in 10 months, or 100% of the enrollment goal within 10 months. Thus, enrollment will be assessed by measuring the percentage of the enrollment goal at the end of 10 months.
Feasibility: Attrition | 10 weeks
  Feasibility will be assessed by examining attrition. Attrition will be measured by the percentage of participants who drop out of the study. The intervention will be considered feasible if >80% of participants complete 6 sessions.
Feasibility: Use of intervention strategies | 10 weeks
  Feasibility will be assessed by examining participants' use of intervention strategies using a novel measure adapted for this study. Participants will be asked how often they have used the strategies presented in the intervention, with responses ranging from 0 ("Not at all") to 5 ("Every day"). Participants will also be asked about how often they have used each individual strategy or skill with responses ranging from 0 ("Not at all") to 4 ("6 or more days/week"). The intervention will be considered feasible if ≥75% of participants report use of intervention skills.
Acceptability: Treatment Acceptability Questionnaire | 10 weeks
  Acceptability will be assessed using the Treatment Acceptability Questionnaire (TAQ). The Treatment Acceptability Questionnaire (TAQ) is a six-item scale assessing whether participants view an intervention as acceptable, ethical, and effective. Items are rated on a 7-point Likert scale (e.g., 1 "very unacceptable" to 7 "very acceptable"). The intervention will be considered acceptable if >80% of participants rate the intervention as >5 out of 7 on the TAQ.
Acceptability: Client Satisfaction Questionnaire | 10 weeks
  Acceptability will be assessed using the Client Satisfaction Questionnaire (CSQ). The CSQ is an 8-item self-report scale to assess participant satisfaction; each item on this scale is scored from 1 to 4, with higher scores indicating higher satisfaction. The intervention will be considered acceptable if >80% of participants rate the intervention as >3 out of 4 on the CSQ.

SECONDARY OUTCOMES:
Change in risk-based knowledge | Baseline, 10 weeks
  Knowledge will be assessed using an item pool developed for the study. Each participant will complete 10 items based on the risk-based education they received. Knowledge will be calculated as the percent of correct items (from 0% to 100%).
Change in symptom severity and interference: menopause symptoms | Baseline, 10 weeks
  Symptom severity and interference will be measured via the Menopause Specific Quality of Life Questionnaire (MENQOL). The 32-item MENQOL assesses the degree of symptom interference in the past week related to four domains: physical symptoms, vasomotor symptoms, psychosocial symptoms, and sexual symptoms. For each symptom that a participant endorses, they will be asked to rate how much they have been bothered by the symptom on a 7-point scale from 0 ("Not at all bothered") to 6 ("Extremely bothered").
Change in symptom severity and interference: anxiety | Baseline, 10 weeks
  Symptom severity and interference will be measured via the PROMIS® Anxiety 8-item Short Form, an 8-item measure assessing symptoms of anxiety in the last week. Participants are asked to respond to items (e.g., "I felt nervous," "I felt tense") using a five-point scale ranging from 1 "never" to 5 "always".
Change in symptom severity and interference: depression | Baseline, 10 weeks
  Symptom severity and interference will be measured via the PROMIS® Depression 8-item Short Form, an 8-item measure assessing symptoms of depression in the last week. Participants are asked to respond to items (e.g., "I felt sad," "I felt helpless") using a five-point scale ranging from 1 "never" to 5 "always."
Change in symptom severity and interference: illness intrusiveness | Baseline, 10 weeks
  Symptom severity and interference will be measured via the Illness Intrusiveness Rating Scale (IIRS). The IIRS assesses the extent to which an illness and/ or its treatments interfere with 13 quality of life domains (e.g., health, diet, work, sex life, active recreation). Items are rated on a 7-point scale from 1 "not very much" to 7 "very much."
Change in decisional conflict | Baseline, 10 weeks
  Decisional conflict related to menopause management will be assessed using the Decisional Conflict Scale (DCS). The DCS is a 16-item measure assessing decisional conflict. The response ranges are on a 5-point Likert scale ranging from strongly agree to strongly disagree. The minimum score is a 0 and the maximum score is 100, with higher scores indicating more decisional conflict.
Change in self-efficacy: decision self-efficacy | Baseline, 10 weeks
  Self-efficacy will be assessed using the Decision Self-Efficacy Scale, an 11-item measure which assesses self-confidence or belief in one's abilities in decision making, including shared decision making. Responses to each item range from 0 (not at all confident) to 4 (very confident).
Change in self-efficacy: self-efficacy for managing symptoms | Baseline, 10 weeks
  Self-efficacy for managing symptoms will be assessed using an 8-item measure in which participants are asked to rate how confident they are that they can manage common symptoms related to menopause. Participants will be asked to rate their confidence in managing symptoms on a 10-point scale from 1 ("Not at all confident") to 10 ("Very confident").
Change in patient activation | Baseline, 10 weeks
  Patient activation will be assessed using the Patient Activation Measure (PAM). The PAM is a 13-item measure used to assess survivors' knowledge, skills, and confidence that are central to managing their health and health care. Patients are asked to rate their agreement with statements about their health and health care on a 4 point scale from "strongly disagree" to "strongly agree." From these response a total PAM score is calculated on a scale of 0-100, with higher scores indicating higher levels of activation.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Shelby, PhD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: Yes